CLINICAL TRIAL: NCT01630512
Title: Mindfulness-Based Cognitive Therapy (MBCT) and Cognitive Behavioral Therapy (CBT) for Depression in Patients With Diabetes: a Randomized Controlled Trial
Brief Title: Mindfulness-Based Cognitive Therapy (MBCT) and Cognitive Behavioral Therapy (CBT) for Depression in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METIS
Record Dates: First submitted 2012-06-15; First posted 2012-06-28 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- MBCT (Experimental)
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — The intervention consists of 8 weekly individual sessions of MBCT. Each session will be administered individually and will last 45 to 60 minutes.
  Arms: MBCT
Behavioral: Cognitive Behavioral Therapy (CBT) — The intervention consists of 8 weekly individual sessions of CBT. Each session will be administered individually and will last 45 to 60 minutes.
  Arms: CBT

SUMMARY:
The purpose of this study is to determine whether mindfulness-based cognitive therapy (MBCT)and cognitive behavioral therapy (CBT)are effective in reducing depressive symptoms in patients with diabetes.

DETAILED DESCRIPTION:
Depression is a common co-morbidity of diabetes, negatively affecting physical performance, glycemic control, adherence to medication, and dietary, and exercise recommendations. Modalities of psychotherapy like cognitive behavioral therapy (CBT) and mindfulness-based cognitive therapy (MBCT) can reduce depressive symptoms in patients with medical conditions. However, proper designed randomized trials assessing and comparing effectiveness of these psychological interventions are rare.

This longitudinal study aims to investigate the effectiveness of CBT and MBCT in reducing depressive symptoms in diabetes patients. Furthermore, potential moderators and mediators of treatment effect will be explored, as well as the role of common factors and treatment integrity.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 1 or 2 for at least three months prior to inclusion
* Written informed consent
* Age ≥ 18 and ≤ 70
* Depressive symptoms as assessed by BDI-II score ≥ 14 (cut-off score indicating the presence of at least mild symptoms of depression)

Exclusion Criteria:

* Not being able to read and write Dutch
* Severe (psychiatric) co-morbidity
* Acute suicidal ideations or behavior
* Pregnancy
* Receiving an alternative psychological treatment during or less than two months prior to starting the participation in the study

Using an antidepressant drug during participation in the present study is allowed, on condition that a patient has been on stable medication regimen for at least two months prior to inclusion in the study, and that no new treatment with an antidepressant is initiated during the course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change in severity of depressive symptoms | change from baseline in severity of depressive symptoms at 3 months, 6 months, and 12 months
  severity of depressive symptoms will be assessed with the Beck Depression Inventory-II

SECONDARY OUTCOMES:
change in diabetes related distress | change from baseline in diabetes related distress at 3 months, 6 months, and 12 months
  diabetes related distress will be measured by the Problem Areas in Diabetes scale (PAID)
change in generalized anxiety | change from baseline in generalized anxiety at 3 months, 6 months, and 12 months
  generalized anxiety will be measured by the Generalised Anxiety Disorder Assessment (GAD 7)
change in well-being | change from baseline in well-being at 3 months, 6 months, and 12 months
  well-being will be measured by the Well-being Index (WHO-5)
change in depressive symptoms | change from baseline in depressive symptoms at 3 months, 6 months, and 12 months
  depressive symptoms will be measured by the 7-Item Hamilton Depression Rating scale (HAM-D7)
change in glycemic control | change from baseline in glycemic control at post-treatment
  glycemic control will be indicated with HbA1c values
intersession changes in mood | change in mood from the beginning of the first session to the beginning of the last session
  intersession changes in mood will be assessed by the Emotion Thermometers Tool (ETT)

CONTACTS AND LOCATIONS:
Overall Officials: Robbert Sanderman, Prof. dr., Study Chair — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

REFERENCES:
- [Derived] Tovote KA, Fleer J, Snippe E, Bas IV, Links TP, Emmelkamp PM, Sanderman R, Schroevers MJ. Cognitive behavioral therapy and mindfulness-based cognitive therapy for depressive symptoms in patients with diabetes: design of a randomized controlled trial. BMC Psychol. 2013 Oct 9;1(1):17. doi: 10.1186/2050-7283-1-17. eCollection 2013. PMID 25566369